CLINICAL TRIAL: NCT00339638
Title: Prediagnostic Markers of Adult T-Cell Leukemia/Lymphoma Among Carriers of Human T-Lymphoma Virus Type I: A Collaborative Study
Brief Title: Study of Adult T-Cell Leukemia/Lymphoma Among Carriers of HTLV-1
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905068; 05-C-N068; NCT00897013 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-05-26

CONDITIONS: Human T-Lymphoma Virus Type I
Keywords: Epidemiology; Risk Prediction; Biomarkers; Nested Case Control

SUMMARY:
This study will identify chemical and protein markers in the blood of people who carry the human T-lymphotropic virus type I (HTLV-I), a virus associated with various pathologies, including an increased risk in adults of a rare and aggressive cancer called adult T cell leukemia/lymphoma (ATL). The study will also examine differences in these markers before and after the onset of ATL.

ATL has been reported in every area where HTLV-1 is common, including the Caribbean and parts of Japan, West Africa, the Middle East, South America, and Pacific Melanesia. Risk factors for the disease are largely unknown and seem to vary among those affected in different endemic regions. People who acquire the infection early in life are thought to be at higher risk than those who are infected later. In Japan, men seem to be at greater risk than women, but the same is not evident among the black population in the Caribbean and Brazil.

Findings from this study will increase understanding of the cause of ATL and identify differences in tumor characteristics and the course of disease across geographical areas.

Study subjects are drawn from among participants in eight studies of HTLV-1 carriers, including the 1) Jamaica Mother-Infant Cohort Study, 2) Jamaica Family Study, 3) Jamaica Food Handlers Study, 4) Miyazaki Cohort Study in Japan, 5) Nagasaki Cohort Study in Japan, 6) Japan Public Health Center-based Prospective Study on Cancer and Cardiovascular Disease, 7) HTLV Outcome Studies in the United States, and 8) GIPH Cohort Study in Brazil.

Stored blood samples previously collected from patients in the above studies who did and did not develop ATL will be analyzed for immunologic and genetic factors.

DETAILED DESCRIPTION:
To characterize molecular markers for risk of adult T-cell leukemia/lymphoma (ATL), whose incidence rate differs greatly across geographic areas, we propose to examine the prevalence and level of viral and host immune response markers as well as the protein expression pattern of 57 subjects who subsequently developed ATL and 171 matched control subjects who participated in various prospective studies of carriers of human T-lymphotropic virus type I (HTLV-I). Informative markers to be studied include provirus load, HTLV-I antibody titer, anti-Tax protein, clonality of HTLV-I infected lymphocytes (viral markers), total immunoglobulin E (IgE), C-reactive protein (CRP), neopterin, soluble CD30, soluble interleukin-2 receptor (sIL2-R), EBV antibody profile (host immune markers), and proteomics. These markers were selected based on the measurability on the majority of specimens, availability of validated assays, relevance to the biology of T-cell malignancies, and has been used in a cross-sectional comparison of HTLV-I carriers and non-carriers from Japan and the Caribbean. We will utilize central laboratory and validated, standard assays for all specimens. The results, unlinked to personal identifiers, will be analyzed using generalized estimating equation. The findings will further our understanding of the etiology of ATL, and of differences in natural history of HTLV-I infection across geographic areas.

While pursuing the same theme of trying to identify host and viral markers associated with ATL, the unique aspect of this proposal is to pool ATL cases, an extremely rare malignancy, from multiple epidemiologic studies through international collaboration, in order to achieve adequate statistical power and to perform valid comparison of tumor characteristics across geographic areas.

ELIGIBILITY:
* INCLUSION CRITERIA:

CASES:

Incident ATL cases will be identified from the various study cohorts. For Jamaica Family Study, in which prevalent cases were enrolled, we will only include cases that occurred among initially unaffected family members. The diagnosis of ATL follows universal criteria for all cohorts. For each case, one prediagnostic specimen will be analyzed. If there are more than one prediagnostic specimens, we will select the earliest drawdate from which both serum/plasma and DNA specimens are available. Whenever available, one postdiagnostic specimen will also be considered for analysis of longitudinal changes in marker levels.

CONTROLS:

Fro each index case, 2 age-, sex-, screen-matched asymptomatic HTLV-I carriers will be selected as controls, from within the same cohort in which the case arose (risk set sampling). For Jamaica Family Study, the control subjects are selected from unrelated subjects (such as spouses or incidental recruit unrelated to the index case) or from one or two population-based studies of unrelated subjects (i.e., food handlers study or mother-infant cohort study). For controls, specimens collected close to the time of pre- and post-diagnostic phlebotomy for the case will be analyzed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2004-12-21; Study Completion 2011-05-26

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Harvard School of Public Health, Boston, Massachusetts
- University of the West Indies, Kingston, Jamaica
- Japan (2):
  - Tokushima University, Tokushima
  - National Cancer Center Research Institute, Toyko

REFERENCES:
- [Background] Manns A, Hisada M, La Grenade L. Human T-lymphotropic virus type I infection. Lancet. 1999 Jun 5;353(9168):1951-8. doi: 10.1016/s0140-6736(98)09460-4. PMID 10371587
- [Background] Uchiyama T, Yodoi J, Sagawa K, Takatsuki K, Uchino H. Adult T-cell leukemia: clinical and hematologic features of 16 cases. Blood. 1977 Sep;50(3):481-92. No abstract available. PMID 301762
- [Background] Yamaguchi K, Seiki M, Yoshida M, Nishimura H, Kawano F, Takatsuki K. The detection of human T cell leukemia virus proviral DNA and its application for classification and diagnosis of T cell malignancy. Blood. 1984 May;63(5):1235-40. PMID 6324929